CLINICAL TRIAL: NCT01858220
Title: Open Prospective Single Center Study for the Determination of Correlation Between Video Capsule Period of Retention in the Stomach and Symptoms of Gastroparesis
Brief Title: IS There a Correlation Between Sypmtoms of Gastroparesis and the Duration of Video Caspule Retention in the Stomach
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Dan Carter, Gastroenterologist, Senior GI Consult, Sheba Medical Center
Other Study IDs: Sheba-9180-2011
Record Dates: First submitted 2013-05-12; First posted 2013-05-21 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Gastroparesis
Keywords: Gastroparesis; Small bowel video capsule; gastric retention
MeSH Terms: conditions — Gastroparesis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Video capsule examinee: Every subject having capsule endoscopy for any indication

SUMMARY:
Gastroparesis is a syndrome characterized by delayed gastric emptying in absence of mechanical obstruction of the stomach. The cardinal symptoms include postprandial fullness (early satiety), nausea, vomiting, and bloating.Capsule endoscopy (CE) has evolved to become a first-line, noninvasive diagnostic technique for the small bowel. CE is now being utilized to assess patients for obscure gastrointestinal bleeding, possible Crohn's disease, celiac disease and small bowel tumors. Capsule endoscopy is preformed in a fasting state, and usually past the pylorus of the stomach into the duodenum after up to 30-40 minutes. The aim of the study is to determine the correlation between gasytoparesis symptoms to duration of capsule retention in the stomach

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Undergoing video capsule endoscopy for any indication

Exclusion Criteria:

-Endoscopic intraduodenal insertion of the capsule -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing small bowel video capsule examination for any indication
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2013-01; Primary Completion 2014-06 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Duration of capsule retention in the stomach | End of capsule examination

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel